CLINICAL TRIAL: NCT00888927
Title: Open-Label, Multi-Center, Dose Escalation Phase 1/2 Study of Anti-CCR4 Monoclonal Antibody KW-0761 as Monotherapy in Subjects With Previously Treated Peripheral T-Cell Lymphoma
Brief Title: Safety Study to Evaluate Monoclonal Antibody KW-0761 in Subjects With Peripheral T-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KW-0761-001
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: T-Cell Lymphoma; PTCL; CTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1 Cohort 1 (Experimental): First course: 0.1 mg/kg once a week over 1 hour for 4 weeks Subsequent courses: 0.1 mg/kg over 1 hour every other week
  Interventions: Biological: KW-0761
- Phase 1 Cohort 2 (Experimental): First course: 0.3 mg/kg once a week over 1 hour for 4 weeks Subsequent courses: 0.3 mg/kg over 1 hour every other week
  Interventions: Biological: KW-0761
- Phase 1 Cohort 3 (Experimental): First course: 1.0 mg/kg once a week over 1 hour for 4 weeks Subsequent courses: 1.0 mg/kg over 1 hour every other week
  Interventions: Biological: KW-0761
- Phase 2 (Experimental): First course: Maximum tolerated dose once a week over 1 hour for 4 weeks Subsequent courses: Maximum tolerated dose over 1 hour every other week
  Interventions: Biological: KW-0761

INTERVENTIONS:
Biological: KW-0761 — The starting dose will be 0.1 mg/kg administered i.v. once every week for four weeks, followed by a 2-week observation period in the first treatment course. Succeeding dose levels will include 0.3 and 1 mg/kg. If a subject has demonstrated an overall CR, may continue on study for up to an additional four infusions beyond CR on an every other week infusion schedule. If a subject experiences a PR or SD, the subject may continue therapy on an every other week infusion schedule until disease progression occurs or other withdrawal criteria are met.

SUMMARY:
This study will determine the maximum dose of KW-0761 administered intravenously that can be given safely in subjects with previously treated peripheral T-cell lymphoma (PTCL) or cutaneous T-cell lymphoma(CTCL)and will see if it is effective in treating the disease.

DETAILED DESCRIPTION:
This Phase 1/2, multicenter, open-label, dose escalation clinical study will enroll up to 47 subjects with previously treated PTCL including CTCL. The study is comprised of a dose escalation phase (Phase 1) and a preliminary assessment of efficacy (Phase 2).

In the dose escalation phase, the starting dose will be 0.1 mg/kg administered i.v. once every week for four weeks, followed by a 2-week observation period in the first treatment course. Succeeding dose levels will include 0.3 and 1 mg/kg. During the first course of treatment if assessments performed at day 29 (end of week 4) indicate that a subject has demonstrated an overall CR, the subject may continue on study for up to an additional four infusions beyond CR on an every other week infusion schedule. Treatment will then be discontinued in order to determine duration of response. If a subject experiences a PR or SD, the subject may continue therapy after consultation between the investigator and the medical monitor on an every other week infusion schedule until disease progression occurs or other withdrawal criteria are met.

ELIGIBILITY:
Inclusion Criteria:

1. histologically/cytologically confirmed diagnosis of PTCL including CTCL (including MF and SS) but excluding ATLL.
2. failed at least one prior systemic therapy for PTCL or CTCL.
3. ECOG PS of <=2 at study entry.
4. >=18 years of age.
5. completed any prior therapy at least four weeks prior to entry; however, patients with rapidly progressive malignant disease may be enrolled prior to this period after discussion with the medical monitor.
6. resolution of all clinically significant toxic effects of prior cancer therapy to grade ≤1 by the NCI-CTCAE, v.3.0 excluding the specifications required in 7 and 8 below.
7. adequate hematological function: absolute neutrophil count>=1,500 cells/uL and platelets >=100,000 cells/uL except in patients with known bone marrow involvement where absolute neutrophil count must be >=1,000 cells/uL and platelets >=75,000 cells/uL.
8. adequate hepatic function: bilirubin ≤ 1.5 times the specific institutional ULN; aspartate transaminase and alanine transaminase each ≤ 2.5 x ULN or ≤ 5.0 x ULN in the presence of known hepatic malignancy.
9. serum creatinine ≤1.5 x ULN or a calculated creatinine clearance >60 mL/min.
10. CTCL subjects previously treated with zanolimumab are eligible provided their CD4+ cell counts have recovered to pre-treatment levels.
11. Subjects with MF and a history of staphylococcus colonization are eligible provided they continue to receive stable doses of prophylactic antibiotics.
12. provided signed informed consent.
13. WOCBP must have a negative pregnancy test within 7 days of receiving study medication.
14. WOCBP must agree to use effective contraception
15. Male subjects must be willing to use an appropriate method of contraception (e.g., condoms) or abstain from sexual intercourse and inform any sexual partners that they must also use a reliable method of contraception during the study.

Exclusion Criteria:

1. has a significant uncontrolled intercurrent illness including, but not limited to: uncontrolled infection requiring antibiotics; clinically significant cardiac disease (class III or IV of the New York Heart Association [NYHA] classification); unstable angina pectoris; angioplasty, stenting, or myocardial infarction within 6 months; uncontrolled hypertension (systolic blood pressure >160 mm Hg, diastolic BP >100 mmHg, found on two consecutive measurements separated by a 1-week period) despite two anti-hypertensive medications; clinically significant cardiac arrhythmia; or uncontrolled diabetes.
2. has known or tests positive for human immunodeficiency virus (HIV), human T-cell leukemia virus (HTLV-1), hepatitis B or hepatitis C.
3. has evidence of central nervous system (CNS) metastasis.
4. has received monoclonal antibodies within 6 weeks of study entry.
5. is pregnant (confirmed by beta human chorionic gonadotrophin [β-HCG]) or lactating.
6. Subjects on any immunomodulatory drug, (other than low dose corticosteroids equivalent to a daily dose of 10 mg of prednisone). Subjects on any immunomodulatory drug within 4 weeks of their first dose of KW-0761 are also excluded.
7. has a psychiatric illness, disability or social situation that would compromise the subject's safety or ability to provide consent, or limit his or her compliance with study requirements.
8. has experienced allergic reactions to monoclonal antibodies or other therapeutic proteins.
9. Subjects with active herpes simplex or herpes zoster. Subjects with a history of herpes zoster who have had an outbreak within the last year will also be excluded. Subjects on prophylaxis for herpes who started taking medication at least 30 days prior to study entry, should continue to take the prescribed medication for the duration of the study.
10. Subjects with known autoimmune diseases. Subjects with Hashimoto's thyroiditis controlled with medication are eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (5):
- United States (5):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford Medical Center, Stanford, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - M.D.Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Duvic M, Pinter-Brown LC, Foss FM, Sokol L, Jorgensen JL, Challagundla P, Dwyer KM, Zhang X, Kurman MR, Ballerini R, Liu L, Kim YH. Phase 1/2 study of mogamulizumab, a defucosylated anti-CCR4 antibody, in previously treated patients with cutaneous T-cell lymphoma. Blood. 2015 Mar 19;125(12):1883-9. doi: 10.1182/blood-2014-09-600924. Epub 2015 Jan 20. PMID 25605368

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Cohort 1: First course: 0.1 mg/kg once a week over 1 hour for 4 weeks Subsequent courses: 0.1 mg/kg over 1 hour every other week
  KW-0761: The starting dose will be 0.1 mg/kg administered i.v. once every week for four weeks, followed by a 2-week observation period in the first treatment course. If a subject has demonstrated an overall CR, may continue on study for up to an additional four infusions beyond CR on an every other week infusion schedule. If a subject experiences a PR or SD, the subject may continue therapy on an every other week infusion schedule until disease progression occurs or other withdrawal criteria are met.
- Phase 1 Cohort 2: First course: 0.3 mg/kg once a week over 1 hour for 4 weeks Subsequent courses: 0.3 mg/kg over 1 hour every other week
  KW-0761: The starting dose will be 0.3 mg/kg administered i.v. once every week for four weeks, followed by a 2-week observation period in the first treatment course. If a subject has demonstrated an overall CR, may continue on study for up to an additional four infusions beyond CR on an every other week infusion schedule. If a subject experiences a PR or SD, the subject may continue therapy on an every other week infusion schedule until disease progression occurs or other withdrawal criteria are met.
- Phase 1 Cohort 3: First course: 1.0 mg/kg once a week over 1 hour for 4 weeks Subsequent courses: 1.0 mg/kg over 1 hour every other week
  KW-0761: The starting dose will be 1.0 mg/kg administered i.v. once every week for four weeks, followed by a 2-week observation period in the first treatment course. If a subject has demonstrated an overall CR, may continue on study for up to an additional four infusions beyond CR on an every other week infusion schedule. If a subject experiences a PR or SD, the subject may continue therapy on an every other week infusion schedule until disease progression occurs or other withdrawal criteria are met.
- Phase 2: First course: Maximum tolerated dose once a week over 1 hour for 4 weeks Subsequent courses: Maximum tolerated dose over 1 hour every other week
  If a subject has demonstrated an overall CR, may continue on study for up to an additional four infusions beyond CR on an every other week infusion schedule. If a subject experiences a PR or SD, the subject may continue therapy on an every other week infusion schedule until disease progression occurs or other withdrawal criteria are met.
Period: Overall Study
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2 | Phase 1 Cohort 3 | Phase 2
Started | 3 | 3 | 3 | 33
Completed | 3 | 3 | 3 | 31
Not Completed | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal of consent | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2 | Phase 1 Cohort 3 | Phase 2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 33 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 12 | 16
  >=65 years | 2 | 2 | 1 | 21 | 26
Age, Continuous [Mean (Full Range); unit: years] | 66 [62 to 68] | 72.3 [64 to 79] | 63.3 [46 to 81] | 66.7 [35 to 85] | 66.8 [35 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 15 | 18
  Male | 3 | 1 | 2 | 18 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black or African American | 1 | 0 | 0 | 2 | 3
  Race/Ethnicity: White/Caucasian, Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Race/Ethnicity: White/Caucasian, Not Hispanic or Latino | 1 | 3 | 3 | 24 | 31
  Race/Ethnicity: White/Caucasian, Not Reported | 0 | 0 | 0 | 4 | 4
  Race/Ethnicity: Other, Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Race/Ethnicity: Not Reported, Not Hispanic or Latino | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 33 | 42

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The objective was to find the maximum tolerated dose (MTD). In the dose escalation phase (Phase 1), the starting dose was 0.1 mg/kg administered intravenously once every week for four weeks, followed by a 2-week observation period in the first treatment course. Succeeding dose levels included 0.3 and 1.0 mg/kg. Standard 3+3 cohorts for safety and DLT detection were utilized. Each cohort consisted of at least three subjects. If Dose-Limiting Toxicity (DLT) was observed in 0/3 subjects, escalation to the next dose level occurred.
Time Frame: 6 weeks
Population: Safety Analysis set - Included all subjects who received at least one dose of KW-0761 (even a partial dose)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2 | Phase 1 Cohort 3 | Phase 2
Number analyzed (Participants) | 3 | 3 | 3 | 33
Participants
  Subjects with any Dose-Limiting Toxicity (DLT) | 0 | 0 | 0 | 0
  Subjects with any treatment emergent adverse event (TEAE) | 3 | 3 | 3 | 32
  Subjects with any treatment-emergent serious adverse event | 0 | 1 | 1 | 8
  Subjects with any TEAE(s) leading to discontinuation | 0 | 1 | 0 | 7

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate was determined based on the response in all compartments (lymph nodes, skin, and viscera) as follows: Complete Response (CR) = complete disappearance of all clinical evidence of disease; Partial Response (PR) = regression of measurable disease; Stable Disease (SD) = failure to attain CR, PR, or PD; Progressive Disease (PD) = PD in any compartment; Relapse = recurrence of disease in prior CR in any compartment.
Time Frame: one year
Population: Efficacy Analysis Set: all subjects who received at least four doses of KW-0761 and had at least one on-study assessment for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2 | Phase 1 Cohort 3 | Phase 2
Number analyzed (Participants) | 3 | 3 | 3 | 30
Participants | 2 | 2 | 1 | 9

ADVERSE EVENTS:
Time Frame: Between the date of first dose and within 30 days after the last dose, up to one year
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2 | Phase 1 Cohort 3 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 2/33
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 8/33
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1 (N=3) | Phase 1 Cohort 2 (N=3) | Phase 1 Cohort 3 (N=3) | Phase 2 (N=33)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1 (N=3) | Phase 1 Cohort 2 (N=3) | Phase 1 Cohort 3 (N=3) | Phase 2 (N=33)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 9 (10)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 9 (12)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (8)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 2 (4) | 1 (1) | 6 (8)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea manuum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (8)
Facial palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 5 (5)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spider vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days